CLINICAL TRIAL: NCT01897363
Title: Hypoglycemia in Prader-Willi Syndrome: A Prospective Study
Brief Title: Hypoglycemia in Prader-Willi Syndrome
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Foundation for Prader-Willi Research (Other)
Responsible Party: Sponsor
Other Study IDs: 59-2013
Record Dates: First submitted 2013-07-08; First posted 2013-07-12 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Prader Willi Syndrome; Hypoglycemia
Keywords: Prader Willi Syndrome; Hypoglycemia; Fasting study
MeSH Terms: conditions — Prader-Willi Syndrome; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants with Prader-Willi Syndrome: Infants between ages 2 to 12 months of age with Prader-Willi Syndrome.
  Interventions: Other: Infants with Prader-Willi Syndrome

INTERVENTIONS:
Other: Infants with Prader-Willi Syndrome — Participants will be admitted to the outpatient clinical research center for IV placement, blood draws from the IV, poking the participants finger to obtain small amounts of blood and monitored 6 hour fast.

SUMMARY:
This project will study whether infants with Prader-Willi Syndrome experience low blood sugars after short periods of fasting. This study will also evaluate metabolic markers in the blood to determine if infants with Prader-Willi Syndrome process energy differently than other children during fasting.

DETAILED DESCRIPTION:
This study will include outpatient admission to the clinical research center for IV placement, blood draws from the IV, poking the participants finger to obtain small amounts of blood and monitored 6 hour fast. A fast is when a person goes without food for a certain period of time. The participant will not be fasted longer than 6 hours.

The participant will arrive to the outpatient clinical research center at approximately 7am. A parent will be expected to stay with the participant at all times. The participant's finger will be poked for blood (requires approximately one drop of blood) soon after arrival to make sure his blood sugar is not already low. If the participant's blood sugar is low on arrival to the Clinical Research Center, additional blood will be drawn through his vein (a little more than half a teaspoon) and he will not have to complete the rest of the study. If his blood glucose is above 60 mg/dl, the participant will be given an opportunity to eat prior to starting the fast. A small tube will be placed in the participant's vein at the beginning of the fast to make additional blood draws easier. 1/10th a teaspoon of blood will be sent for cortisol testing when the IV is placed. Cortisol is a hormone that is important for control of blood sugar. In addition, the participant's finger will be pricked every hour for blood to monitor his blood sugar by bedside meter. Each finger prick will require approximately one to two drops of blood. A test to look at fat breakdown (ketones) will sometimes be checked using the same blood obtained when pricking the finger to check blood sugar. If a blood sugar of less than 70 mg/dl is found, blood sugars will be checked by finger prick every 30 minutes instead of every hour. If finger prick blood glucose is less than 65 mg/dl, blood will be collected and sent to the clinical research center lab to make sure that the true blood sugar reading is not lower than what is seen on the bedside meter (requires approximately 1/10 teaspoon of blood). If a blood sugar of less than 60 mg/dl is found, the fast will end and blood will be collected through the IV line (small tube placed through the vein). The participant will be monitored by a nurse during the fast. She will check his blood pressure, pulse and respiratory rate periodically to make sure he is comfortable. After final blood collection, the participant will be allowed to feed normally and his IV will be removed. During the entire study, we expect to collect at least ¾ of a teaspoon of blood from the participant. No more than 1.2 teaspoons of blood will be collected from the participant during this entire study.

If a blood sugar less than 60 mg/dl is found at any time, blood will be drawn from a vein in the participant's arm and the study will end. He will then be allowed to eat. If he has a low blood sugar and is unable to feed the way he normally does, sugar water/gel may be given by mouth or sugar water may be given by the tube placed in his vein. If the participant normally is fed by a tube placed in his stomach, sugar water may be given through this tube.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Prader-Willi Syndrome
* Between ages 2-12 months of age
* Determined to be in nutritional phase 1a by clinical assessment

Exclusion Criteria:

* Treatment with growth hormone

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with Prader-Willi Syndrome who have not yet started growth hormone therapy
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Presence of hypoglycemia | During 6 hours of fasting
  We will determine whether fasting occurs within 6 hours of fasting in infants with Prader-Willi Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Miller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States